CLINICAL TRIAL: NCT00676741
Title: Observational Study on Evaluation of Glycaemic Control in Patients Using a Modern Insulin - NovoRapid® (Insulin Aspart), NovoMix® 30 (Biphasic Insulin Aspart) or Levemir® (Insulin Detemir) - for Treatment of Diabetes Mellitus
Brief Title: Observational Study on Blood Glucose Control in Patients With Diabetes Using Modern Insulin
Acronym: COMMIT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: BIASP-3516
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A
  Interventions: Drug: insulin aspart
- B
  Interventions: Drug: biphasic insulin aspart 30
- C
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin aspart — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: NovoRapid®
  Groups: A
Drug: biphasic insulin aspart 30 — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Groups: B
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Groups: C

SUMMARY:
The study is conducted in Europe. The aim of this observational study is to evaluate the blood glucose control in patients using a modern insulin: NovoRapid®, NovoMix® 30 or Levemir® for the treatment type 2 diabetes.

Full acronym for this study: COMMIT - CLEAN SWITCH

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes
* Patients treated with human soluble insulin, NPH insulin or premixed human insulin
* Patients willing to sign informed consent
* Selection of study participants at the discretion of the physician

Exclusion Criteria:

* Subjects currently being treated with insulin aspart, insulin detemir or biphasic insulin aspart 30
* Subjects who were previously enrolled in this study
* Subjects with a hypersensitivity to insulin aspart, insulin detemir or biphasic insulin aspart 30 or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes type 2
Sampling Method: Non-Probability Sample
Enrollment: 3809 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Metabolic control measured as HbA1c | for the duration of the study

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c below 7.0% and below or equal 6.5% | after 12 weeks and 24 weeks
Change in FPG (glucose variability) | after 12 weeks and 24 weeks
Change in PPG (postprandial control) | after 12 weeks and 24 weeks
Change in insulin dose and number of injections | after 12 weeks and 24 weeks
Change in oral antidiabetic drug therapy | after 12 weeks and 24 weeks
Change in body weight | after 12 weeks and 24 weeks
Change in number of hypoglycaemic events during 4 weeks proceeding routine visits | after 12 weeks and 24 weeks
Number of adverse drug reactions (ADR) | after 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com